CLINICAL TRIAL: NCT05754892
Title: Positioning of Molecular Markers in Clinical Routine for the Management of Patients With Adrenal Cancers/Tumors (COMETE-CARE)
Acronym: COMETE-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210350; 2022-A00663-40 (Other: ID-RCB Number)
Record Dates: First submitted 2022-12-26; First posted 2023-03-06 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Adrenal
Keywords: biological markers; genomics
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ACC (Other): These patients will be followed up and proposed a search for targetable molecular alterations
  Interventions: Other: Blood sample; Other: Urine sample; Other: Tumor sample
- Patients with MPP (Other): These patients will be followed up and proposed a search for targetable molecular alterations
  Interventions: Other: Blood sample; Other: Urine sample; Other: Tumor sample

INTERVENTIONS:
Other: Blood sample — For patients with ACC : blood (30ml) sampling before surgery and every 3 months during 3 years after surgery for biobanking For patients with MPP : blood (30ml) sampling before surgery and every 6 to 12 months for MPP during 3 years after surgery for biobanking
Other: Urine sample — For patients with ACC : urine sampling before surgery and every 3 months during 3 years after surgery for biobanking For patients with MPP : urine sampling before surgery and every 6 to 12 months for MPP during 3 years after surgery for biobanking
Other: Tumor sample — For patients with ACC and patients with MPP : tumor sample during surgery

SUMMARY:
The adrenal cancer research network "COMETE" is federating French research on rare adrenal cancers. COMETE achieved major breakthroughs in the molecular characterization of adrenocortical carcinomas (ACC) and malignant pheochromocytomas/paragangliomas (MPP). Recently, COMETE successfully derived potential biomarkers for prognosis, theranostic and follow-up. Those biomarkers have been retrospectively validated. However the benefit for patients in real life conditions is not yet established.

* Main objective : to implement COMETE biomarkers as a routine standard of care for adrenal cancer.
* The primary end point is double :

  * Proportion of biomarkers results provided within 3 months after surgery,
  * The proportion of "informative" biomarkers, corresponding to markers passing quality controls and returning a value that is not in the grey zone of the measure.
* Secondary objective : to estimate the impact of COMETE biomarkers on patients management.
* Secondary endpoints :

  * Proportion of patients with discrepant clinical and molecular markers ; for discrepancies, proportion of decisions impacted by biomarkers results
  * Proportion of high risk patients for whom an actionable molecular target was identified
  * Predictive value (positive and negative) of biomarkers to detect recurrences
  * Molecular signatures of "extraordinary responders" to treatments (corresponding to the exceptional RECIST complete response, or to the >80% tumor reduction sutained for >6months)

DETAILED DESCRIPTION:
* Adult patients with a malignant adrenal tumor before initial surgery are proposed to participate to the study.
* Initial clinical management following current guidelines is applied, including clinical and morphological evaluation, hormone assays and adrenal surgery. A tumor sample from initial surgery , and a blood sample and a urine sample collected before surgery are included in the current research protocol. These samples are used to run prognostic molecular measurements, in order to classify patients as "low" or "high risk" of recurrence. For ACC samples, paraffin tumor samples will be sent to a centralized pathology facility, where 3' RNA sequencing will be performed on tumor RNA to classify tumors into previously established C1A/C1B prognostic classification. Circulating levels of miRNAs will be assayed from blood samples collected before surgery and used to classify tumors into prognostic categories as previously reported. Urine and plasma steroids profiles will be established using mass spectrometry to classify tumors into prognostic categories as previously reported. For MPP, molecular assays will include somatic genotyping, methylation assays and immunochemistry for the known recurrently altered genes, and used to classify tumors into prognostic categories as previously reported. These molecular results are returned by 3 months after surgery
* Patients follow-up is then performed following current guidelines, with repeated visits (each ~3 months for ACC and ~6 months for MPP), including clinical, morphological evaluation, and hormone assays. A blood and a urine sample will also be collected for the current research protocol. These samples will be used to run molecular measurements aiming at identifying early recurrence. For ACC, circulating levels of miRNAs and urine and plasma steroids profiles will be measured every 3 months to classify tumors into prognostic categories as previously reported. For MPP, circulating levels of miRNAs will be measured every 6 months to classify tumors into prognostic categories as previously reported
* For patients at high risk of recurrence, a molecular target will be searched by an extended genomic analysis of the tumor (exome sequencing and RNA sequencing), in search for molecular targets that may orient future treatments, if the disease recurs.

ELIGIBILITY:
Inclusion Criteria

* Patients 18 years of age and older
* Patients with an adrenal tumor who will be operated of a potentially malignant adrenocortical carcinoma (ACC) or pheochromocytoma or paraganglioma (MPP) (any stage, any secretion)
* Patients affiliated with a social security regime
* Patients who have signed an informed consent

Exclusion Criteria

* Vulnerable populations : minors, pregnant or breastfeeding women, protected adults
* Patients on AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Baseline biomarkers results | Within 3 months after surgery
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after initial surgery

SECONDARY OUTCOMES:
M3 biomarkers results | During follow-up (month 6)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M6 follow-up visit
M6 biomarkers results | During follow-up (month 9)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M9 follow-up visit
M9 biomarkers results | During follow-up (month 12)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M12 follow-up visit
M12 biomarkers results | During follow-up (month 15)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M15 follow-up visit
M15 biomarkers results | During follow-up (month 18)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M18 follow-up visit
M18 biomarkers results | During follow-up (month 21)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M21 follow-up visit
M21 biomarkers results | During follow-up (month 24)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M24 follow-up visit
M24 biomarkers results | During follow-up (month 27)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M27 follow-up visit
M27 biomarkers results | During follow-up (month 30)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M30 follow-up visit
M30 biomarkers results | During follow-up (month 33)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M33 follow-up visit
M33 biomarkers results | During follow-up (month 36)
  Proportion of biomarkers and of informative biomarkers returned to physicians within 3 months after M36 follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Anne JOUINOT, Dr, Study Director — APHP
Locations (1):
- GH Paris Centre, Assistance Publique - Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Assie G, Jouinot A, Fassnacht M, Libe R, Garinet S, Jacob L, Hamzaoui N, Neou M, Sakat J, de La Villeon B, Perlemoine K, Ragazzon B, Sibony M, Tissier F, Gaujoux S, Dousset B, Sbiera S, Ronchi CL, Kroiss M, Korpershoek E, De Krijger R, Waldmann J, Quinkler M, Haissaguerre M, Tabarin A, Chabre O, Luconi M, Mannelli M, Groussin L, Bertagna X, Baudin E, Amar L, Coste J, Beuschlein F, Bertherat J. Value of Molecular Classification for Prognostic Assessment of Adrenocortical Carcinoma. JAMA Oncol. 2019 Oct 1;5(10):1440-1447. doi: 10.1001/jamaoncol.2019.1558. PMID 31294750
- [Background] Lenders JWM, Kerstens MN, Amar L, Prejbisz A, Robledo M, Taieb D, Pacak K, Crona J, Zelinka T, Mannelli M, Deutschbein T, Timmers HJLM, Castinetti F, Dralle H, Widimsky J, Gimenez-Roqueplo AP, Eisenhofer G. Genetics, diagnosis, management and future directions of research of phaeochromocytoma and paraganglioma: a position statement and consensus of the Working Group on Endocrine Hypertension of the European Society of Hypertension. J Hypertens. 2020 Aug;38(8):1443-1456. doi: 10.1097/HJH.0000000000002438. PMID 32412940
- [Background] Jouinot A, Lippert J, Sibony M, Violon F, Jeanpierre L, De Murat D, Armignacco R, Septier A, Perlemoine K, Letourneur F, Izac B, Ragazzon B, Leroy K, Pasmant E, North MO, Gaujoux S, Dousset B, Groussin L, Libe R, Terris B, Fassnacht M, Ronchi CL, Bertherat J, Assie G. Transcriptome in paraffin samples for the diagnosis and prognosis of adrenocortical carcinoma. Eur J Endocrinol. 2022 Apr 21;186(6):607-617. doi: 10.1530/EJE-21-1228. PMID 35266879
- [Background] Chabre O, Libe R, Assie G, Barreau O, Bertherat J, Bertagna X, Feige JJ, Cherradi N. Serum miR-483-5p and miR-195 are predictive of recurrence risk in adrenocortical cancer patients. Endocr Relat Cancer. 2013 Jul 5;20(4):579-94. doi: 10.1530/ERC-13-0051. Print 2013 Aug. PMID 23756429
- [Background] Bancos I, Taylor AE, Chortis V, Sitch AJ, Jenkinson C, Davidge-Pitts CJ, Lang K, Tsagarakis S, Macech M, Riester A, Deutschbein T, Pupovac ID, Kienitz T, Prete A, Papathomas TG, Gilligan LC, Bancos C, Reimondo G, Haissaguerre M, Marina L, Grytaas MA, Sajwani A, Langton K, Ivison HE, Shackleton CHL, Erickson D, Asia M, Palimeri S, Kondracka A, Spyroglou A, Ronchi CL, Simunov B, Delivanis DA, Sutcliffe RP, Tsirou I, Bednarczuk T, Reincke M, Burger-Stritt S, Feelders RA, Canu L, Haak HR, Eisenhofer G, Dennedy MC, Ueland GA, Ivovic M, Tabarin A, Terzolo M, Quinkler M, Kastelan D, Fassnacht M, Beuschlein F, Ambroziak U, Vassiliadi DA, O'Reilly MW, Young WF Jr, Biehl M, Deeks JJ, Arlt W; ENSAT EURINE-ACT Investigators. Urine steroid metabolomics for the differential diagnosis of adrenal incidentalomas in the EURINE-ACT study: a prospective test validation study. Lancet Diabetes Endocrinol. 2020 Sep;8(9):773-781. doi: 10.1016/S2213-8587(20)30218-7. Epub 2020 Jul 23. PMID 32711725